CLINICAL TRIAL: NCT02136329
Title: A Phase I Study to Determine the Pharmacokinetic Profile, Safety and Tolerability of Sildenafil (REVATIO®) in Cardiac Surgery
Brief Title: A Study to Determine the Pharmacokinetic Profile, Safety and Tolerability of Sildenafil (REVATIO®) in Cardiac Surgery
Acronym: Revaki-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Leicester (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0359
Record Dates: First submitted 2014-05-06; First posted 2014-05-13 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2014-12

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sildenafil (Experimental): All subjects in groups 1-6 will receive SIldenafil but in escalating doses.
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Sildenafil — The active study drug, Revatio®, is the citrate salt of sildenafil, a selective inhibitor of cyclic guanosine monophosphate (cGMP)-specific phosphodiesterase type-5 (PDE5). Sildenafil citrate is designated chemically as 1-[[3-(6,7-dihydro-1-methyl-7-oxo-3-propyl-1H-pyrazolo [4,3-d] pyrimidin-5-yl)-4-ethoxyphenyl] sulfonyl]-4-methylpiperazine citrate.
  The active study medication is supplied in single use glass vials and as a clear, colourless, sterile, ready-to-use solution containing 10 mg (12.5 mL) of sildenafil. Each mL of solution contains 1.124 mg sildenafil citrate, 50.5 mg dextrose and water for injection.
  Sildenafil is manufactured under Good Manufacturing Practice (EU-GMP) by Pfizer Inc
  Other Names: REVATIO®

SUMMARY:
The objectives of the study are the following:

* To evaluate the pharmacokinetic profile of Sildenafil in cardiac surgery patients at risk of acute kidney injury
* To determine the safety and tolerability of Sildenafil in cardiac surgery patients at risk of acute kidney injury

DETAILED DESCRIPTION:
Acute kidney injury occurs in up to one third of all patients following cardiac surgery. It is manifested by an acute decline in kidney function and results in significant increases in postoperative complications as well as an almost fourfold increase in the risk of postoperative death. Our understanding of the underlying processes is poor and recent systematic reviews have concluded that there is no effective treatment.

Experimental studies have demonstrated that preservation of endogenous Nitric Oxide (NO) bioavailability is reno-protective in response to a variety of injurious stimuli. Endogenous NO activity is increased by administration of the phosphodiesterase type 5 (PDE-5) inhibitor sildenafil citrate. This is used clinically in the treatment of erectile dysfunction (Viagra®, Pfizer) and more recently, pulmonary hypertension and acute right ventricular failure (Revatio®, Pfizer). We have developed a preclinical swine model of extracorporeal circulation (cardiopulmonary bypass) mediated acute kidney injury that shows significant homology to that which occurs in post cardiac surgery patients. Administration of intravenous sildenafil prevents acute kidney injury in this model in association with an increase in NO bioavailability. There is a recognized clinical need for developing prevention and treatment strategies for AKI and results obtained in this preclinical study indicate that Sildenafil is suitable for further development as a potential prevention strategy for post cardiac surgery AKI.

Prior to conducting a safety and efficacy trial however we intend to first establish a dose of Sildenafil that is tolerated by cardiac surgery patients and compare the pharmacokinetics of this dose to the effective dose identified in our preclinical work. We therefore propose to evaluate the pharmacokinetic profile, safety and tolerability of sildenafil in 36 patients undergoing cardiac surgery, in an open label, dose escalation Phase I study. This study will inform the design of a subsequent randomized Phase IIb trial that will determine efficacy and safety

ELIGIBILITY:
Inclusion Criteria:

1. Adult cardiac surgery patients (>18 years) undergoing cardiac surgery with moderately hypothermic CPB (32-34°C) and blood cardioplegia
2. Identified as representing a high risk group for acute kidney injury using a modified risk score based on the variables of Age, Sex, BMI, Smoking Status, NHYA class, Previous Operations, Peripheral Vascular Disease, Diabetes, Hypertension, Pre-operative Haemoglobin level, Pre-operative eGFR, Operative Priority, Operation Type, Ejection Fraction and Presence of Pre-Operative Critical Events.
3. Female subjects of childbearing potential are not to be pregnant (to be confirmed by urine human chorionic gonadotropin pregnancy test prior to dosing). Women are considered not to be of childbearing potential if they have been surgically sterilised (eg, tubal ligation, oophorectomy or hysterectomy) or are postmenopausal (defined as serum follicle-stimulating hormone level of ≥30 IU/mL) in the absence of hormone replacement therapy and complete absence of menses for at least 24 consecutive months.

Exclusion Criteria:

1. Emergency or salvage procedure
2. Ejection fraction <30%
3. CKD Stage 5, defined as eGFR<15ml/min or renal replacement therapy.
4. Administration of potent CYP 3A4 inhibitors within 1 month prior to study participation (e.g. HIV protease inhibitors, imidazole antifungals and erythromycin, please see Appendix 1 for a full list of prohibited medications).
5. Administration of nitrate medicines (e.g. glyceryl trinitrate within 24 hours of surgery.
6. Any ongoing malignancy, or prior malignancy that currently requires treatment.
7. Patients allergic to any other PDE-5 Inhibitor
8. Patients who are participating in another interventional clinical study

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve and Plasma Concentration of Sildenafil | 48 Hours
  There will be Pharmacokinetic sample collection pre and post dose to look at plasma concentration of sildenafil. Sample collection timepoints are post dose at 10 mins, 15 mins, 30 mns, 45 mins 2 hours, 4 hours, 12 hours, 24 hours and 48 hours.

SECONDARY OUTCOMES:
Serum creatinine and Biochemical markers of AKI | 5 Days
  Serum creatinine measured from blood samples collected pre-operatively and at 6 hours, 24 hours, 48 hours and 96 hours after the operation.
  Biochemical markers of acute kidney injury measured in urine pre-operatively, 0mins, 6 houts, 24 hours and 48 hours.

OTHER OUTCOMES:
Adverse Events | 6 Weeks
  Adverse Events will be captured from from time of consent to 6 weeks post operation

CONTACTS AND LOCATIONS:
Overall Officials: Gavin Murphy, Prof, Principal Investigator — University of Leicester
Locations (1):
- Department of Cardiovascular Sciences., Leicester, Leicestershire, United Kingdom